CLINICAL TRIAL: NCT05659264
Title: A Phase 1, Adaptive, Open-Label, Single Ascending Dose to Single-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of mRNA-0184 in Participants With Chronic Heart Failure
Brief Title: A Study to Evaluate the Safety of mRNA-0184 in Participants With Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: mRNA-0184-P101; 2022-000784-46 (EudraCT Number)
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Chronic Heart Failure
Keywords: Single ascending dose; Multiple ascending dose; mRNA-0184; Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The single ascending dose (SAD) stage of this study is open-label and the multiple ascending dose (MAD) stage of this study is single-blind and placebo-controlled.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAD Stage: mRNA-0184 (Experimental): Participants will receive a single dose of mRNA-0184.
  Interventions: Drug: mRNA-0184
- MAD Stage: mRNA-0184 (Experimental): Participants will receive up to 4 doses of mRNA-0184 administered over a treatment period of up to 16 weeks.
  Interventions: Drug: mRNA-0184
- MAD Stage: Placebo (Placebo Comparator): Participants will receive placebo matching to mRNA-0184 administered over a treatment period of up to 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mRNA-0184 — mRNA-0184 dispersion for intravenous (IV) infusion
  Arms: MAD Stage: mRNA-0184; SAD Stage: mRNA-0184
Drug: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: MAD Stage: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of single and multiple doses at escalating dose levels of mRNA-0184.

DETAILED DESCRIPTION:
The study includes a SAD stage and MAD stage; the stages of SAD and MAD may overlap. The SAD stage will begin first, and data from this stage will inform decisions about dose levels in subsequent SAD cohorts and in the MAD stage.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of heart failure (HF) based on medical records.
* Left ventricular ejection fraction (LVEF) ≥ 35% and < 50% at Screening, or documented within the 3 months before Screening, measured by transthoracic echocardiogram (TTE) or cardiac magnetic resonance imaging (MRI).
* New York Heart Association (NYHA) HF Class I or II.
* On a stable regimen of cardiovascular medication(s) for a duration of at least 4 weeks before Screening.

Key Exclusion Criteria:

* Hospitalized for cardiovascular causes within 3 months before Screening.
* Decompensated HF, acute myocarditis, hypertrophic and/or restrictive/constrictive cardiomyopathy, or moderate or severe valvular heart disease (as classified by echocardiography) at Screening or within the 3 months before Screening. Moderate tricuspid regurgitation is not exclusionary. Congenital heart disease as the primary etiology for heart failure will be excluded.
* Symptoms of angina pectoris at Screening.
* Severe obstructive or restrictive pulmonary pathology, including chronic obstructive pulmonary disease Gold Stage III or IV, current use of oxygen therapy, or Group 1, 3, 4, or 5 pulmonary hypertension. Group 2 pulmonary hypertension is not exclusionary.
* History of sustained ventricular tachycardia or atrial fibrillation/atrial flutter with a ventricular response ≥ 110 beats per minute (bpm) at the time of Screening.
* History of hypersensitivity to any components of the investigational product (IP).
* Participant has received or is expected to receive a COVID-19 vaccination within 7 days of the planned date of IP administration.
* For SAD cohort participants to be rolled over into the MAD stage, have experienced a dose-limiting toxicity (DLT) in a SAD cohort.
* Participation in another clinical study of another IP within 30 days before Screening or within 5 terminal elimination half-lives of the IP, whichever is longer.
* Any other clinically significant medical condition that, in the Investigator's opinion, could interfere with the interpretation of study results or limit the participant's participation in the study, including poorly controlled diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Baseline up to Day 296

SECONDARY OUTCOMES:
Serum Concentrations of mRNA Encoding Relaxin-2-variable Light Chain Kappa (Rel2- vlk mRNA) | Day 1 (within 60 minutes predose) up to Day 183
Maximum Observed Plasma Concentration (Cmax) of Rel2-vlk mRNA | Day 1 (within 60 minutes predose) up to Day 183
Area Under the Curve From Time 0 to Time t (AUC0-t) of Rel2-vlk mRNA | Day 1 (within 60 minutes predose) up to Day 183
Serum Concentrations of Relaxin-2-variable Light Chain Kappa (Rel2- vlk) Protein | Day 1 (within 60 minutes predose) up to Day 183
Maximum Observed Effect (Emax) of Rel2- vlk Protein | Day 1 (within 60 minutes predose) up to Day 183
Area Under the Effect-Time Curve (AUEC) of Rel2-vlk Protein | Day 1 (within 60 minutes predose) up to Day 183
Number of Participants With Anti-polyethylene glycol (PEG) Antibodies | Baseline up to Day 183
Number of Participants With anti-Rel2-vlk Protein Antibodies | Baseline up to Day 183

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - Cardiology PC, Birmingham, Alabama
  - University of Alabama at Birmingham: The Kirklin Clinic, Birmingham, Alabama
  - University of Florida, Gainesville, Florida
  - Jacksonville Center For Clinical Research - ERN - PPDS, Jacksonville, Florida
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan, Greater Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Gornoslaskie Centrum Medyczne im. prof. Leszka Gieca Slasiego Uniwersytetu Medycznego w Katowicach, Katowice, Silesian Voivodeship
- United Kingdom (5):
  - Ninewells Hospital & Medical School, Dundee, Angus
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - University College Hospital, London, City of London
  - Derriford Hospital, Plymouth, Devon
  - The Royal Liverpool University Hospital, Liverpool